CLINICAL TRIAL: NCT06618612
Title: A Multicenter, Prospective, Randomized Controlled Modified Platform Trial Assessing the Efficacy of a Purified Native Type 1 Collagen Extracellular Matrix With Polyhexamethylene Biguanide Antimicrobial (PCMP) and Standard of Care Versus Standard of Care Alone in the Management of Nonhealing Diabetic Foot Ulcers
Brief Title: A Study to Evaluate the Efficacy of a Purified Native Type 1 Collagen Extracellular Matrix With Polyhexamethylene Biguanide Antimicrobial (PCMP) and Standard of Care Versus Standard of Care Alone in the Management of Nonhealing Diabetic Foot Ulcers
Acronym: PREPARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Organogenesis (Industry)
Collaborators: Serena Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OI-24001
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Foot Ulcer
Keywords: DFU; Chronic Diabetic Foot Ulcer; Non-healing DFU
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Standard of Care (Other): Standard of Care (SOC)
  Interventions: Other: Standard of Care
- PuraPly AM + SOC (Active Comparator): PuraPly Antimicrobial Wound Matrix along with standard of care
  Interventions: Other: Standard of Care; Device: PuraPly AM
- PuraPly XT + SOC (Active Comparator): PuraPly Antimicrobial XT Wound Matrix along with standard of care
  Interventions: Other: Standard of Care; Device: PuraPly XT

INTERVENTIONS:
Other: Standard of Care — Standard of Care (SOC) includes, but is not limited to, surgical debridement, aggressive infection management, offloading, and maintenance of appropriate cleansing at the time of each dressing change.
Device: PuraPly AM — PuraPly Antimicrobial Wound Matrix is a 2-layer cross-linked extracellular matrix (PCMP) scaffolding that consists of a collagen sheet coated with 0.1% polyhexamethylenebiguanide hydrochloride (PHMB)
  Arms: PuraPly AM + SOC
Device: PuraPly XT — PuraPly Antimicrobial XT Wound Matrix is a 5- layer cross-linked extracellular matrix (PCMP) scaffolding that consists of a collagen sheet coated with 0.1% polyhexamethylenebiguanide hydrochloride (PHMB)
  Arms: PuraPly XT + SOC

SUMMARY:
This prospective, multi-center, randomized, controlled modified platform Trial compares Purified Native Type 1 Collagen Extracellular Matrix with Polyhexamethylene Biguanide Antimicrobial (PCMP) and Standard of Care versus Standard of Care Alone in subjects with chronic DFUs.

DETAILED DESCRIPTION:
At least 170 subjects with a chronic DFU will be randomized 1.4:1:1 to the SOC group, PuraPly AM + SOC, or PuraPly XT + SOC.

Following screening and randomization, subjects shall be seen weekly for up to 12 weeks. For subjects that heal, a healing confirmation visit shall occur two weeks later to confirm maintenance of complete wound closure.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age or older.
2. Diagnosis of type 1 or 2 Diabetes mellitus.
3. At enrollment, target ulcer with a minimum surface area of 1.0 cm2
4. The target ulcer must have been present for a minimum of 4 weeks
5. The target ulcer must be located on the foot with at least 50% of the ulcer below the malleolus.
6. The target ulcer must be Wagner 1 or 2 grade
7. The affected limb must have adequate perfusion confirmed by vascular assessment.
8. If the potential subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
9. Target ulcers located on the plantar aspect of the foot must be offloaded for at least 14 days prior to enrollment.
10. The potential subject must consent to using the prescribed offloading method for the duration of the study.
11. The potential subject must agree to attend the weekly study visits required by the protocol.
12. The potential subject must be willing and able to participate in the informed consent process.

Exclusion Criteria:

1. The potential subject is known to have a life expectancy of < 6 months.
2. The potential subject's target ulcer is not secondary to diabetes.
3. The target ulcer is infected or there is cellulitis in the surrounding skin.
4. The target ulcer exposes tendon or bone.
5. There is evidence of osteomyelitis
6. There is an infection in the target ulcer or in a remote location that requires systemic antibiotic therapy.
7. The potential subject is receiving immunosuppressants or cytotoxic chemotherapy or is taking medications that the PI believes will interfere with wound healing.
8. The potential subject is taking hydroxyurea.
9. The potential subject has applied topical steroids to the ulcer surface within one month of initial screening.
10. The potential subject with a previous partial amputation on the affected foot that results in a deformity that impedes proper offloading of the target ulcer.
11. The potential subject has a controlled glycated hemoglobin (HbA1c) within 3 months of the initial screening visit.
12. The potential subject has an acute Charcot foot, or an inactive Charcot foot, which impedes proper offloading of the target ulcer.
13. Women who are pregnant or considering becoming pregnant within the next 6 months.
14. The potential subject has end stage renal disease requiring dialysis.
15. Participation in a clinical trial involving treatment with an investigational product within the previous 30 days.
16. A potential subject who, in the opinion of the investigator, has a medical or psychological condition that may interfere with study assessments.
17. The potential subject was treated with hyperbaric oxygen therapy (HBOT) or a Cellular, Acellular, Matrix-like Product (CAMP) in the 30 days prior to the initial screening visit.
18. The potential subject has a malnutrition indicator score <17 as measured on the Mini Nutritional Assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-08-19 (Estimated); Study Completion 2026-11-19 (Estimated)

PRIMARY OUTCOMES:
Determine the efficacy of multiple Polyhexamethylene Biguanide Antimicrobial (PCMPs) plus SOC versus SOC alone in achieving complete closure | 12 weeks
  The percentage of target ulcers achieving complete wound closure in 12 weeks

SECONDARY OUTCOMES:
Time to closure for the target ulcer. | 12 weeks
Percentage wound area reduction from Treatment Visit-1 to Treatment Visit-13 | 12 weeks
The number of adverse events. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maribel Henao, Study Director — Organogenesis
Locations (1):
- Kent State University, College of Podiatric Medicine, Clevland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No